CLINICAL TRIAL: NCT07111819
Title: Cervical Cancer Screening Using Self-sampling Approach: Validation of Human Papillomavirus Self-sampling Kits Among Kazakhstani Women
Brief Title: Cervical Cancer Screening Via Self-sampling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazarbayev University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AP26194759
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer Screening
Keywords: Cervical cancer prevention; HPV; Cervical cancer screening; HPV self-sampling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Validation of self-sampling devices (Other)
  Interventions: Behavioral: Self-sampling acceptance

INTERVENTIONS:
Behavioral: Self-sampling acceptance — Cervical self-sampling devices will be distributed among the study participants followed by survey on the devices acceptance

SUMMARY:
Prevention of cervical cancer is one of the priority areas of the Comprehensive Plan to Combat Cancer in the Republic of Kazakhstan for 2023-2027. High-risk human papillomavirus (HR-HPV) infections cause a wide variety of benign and malignant conditions, including cervical cancer. More than 90% of cervical cancer cases are attributed to HR-HPV infections, with HPV-16 and HPV-18 being reported to cause 70-75% of cases. At the present time, cervical cancer remains the fourth most prevalent cancer among women worldwide. Moreover, the majority of cervical cancer cases (90%) occur in low- and middle-income countries (LMICs), where cervical cancer remains the leading cause of death from cancer. Each year, the number of cervical cancer cases is dynamically increasing globally. Between 2000 and 2020 the absolute number of cervical cancer cases increased from 471 000 to 600 000. In 2020, there were around 350,000 deaths from cervical cancer. Moreover, by 2030 it is estimated that the number of new cervical cancer cases will reach 700 000, and the annual number of deaths will reach 400 000. Therefore, given such a significant annual increase in the number of cases and deaths, the elimination of cervical cancer is a global public health challenge.

The prevalence of HPV infection in Kazakhstan is high, around 39% among women attending gynecological clinics. Consequently, the cervical cancer incidence in Kazakhstan has increased over the past decade, and cervical cancer is the second leading cancer type among women in the country. Moreover, among Central Asian countries, Kazakhstan has the second-highest incidence rate of cervical cancer. The cervical cancer screening program is covered by the government and utilizes Papanicolaou test (Pap-test) performed by gynecologists in outpatient clinics all over the country. However, the screening coverage was reported to be low, covering only around 46% of the eligible population, and does not reach the demand level of 70% suggested by the World Health Organization (WHO). Furthermore, the national HPV vaccination program has just started in September 2024 and could contribute to the reduction of cervical cancer incidence only in the coming 10 years when the effect of vaccination will have an impact on the decrease of HPV prevalence in the country. A proper cervical cancer screening and screening coverage play a crucial role in cervical cancer prevention and control. Thus, there are many factors found to have an impact on overall screening behavior among Kazakhstani women and the increasing incidence of cervical cancer in the country. However, the current screening practices do not show high efficacy due to low coverage and general low sensitivity of the method used. These factors result in growing cervical cancer incidence in Kazakhstan. Thus, there is an emergent need to improve the screening process by introducing novel and reliable methods of screening. Cervical self-sampling could potentially improve the screening coverage; however, the approach should be validated to prove its effectiveness in the Kazakhstani cultural setting before introduction to the healthcare system.

DETAILED DESCRIPTION:
Study subjects and sample size. The study will be performed in the Nazarbayev University School of Medicine (NUSOM) in collaboration with other local medical universities and institutions.

This will be a cross-sectional study involving women attending outpatient clinics in Kazakhstani major cities, who will be recruited into the study to validate the HPV self-sampling kits. The project timeline is - January 2025-December 2027. We plan to invite 1000 women for a validation study: all women will complete a questionnaire after self-collection of a smear using kits.

Inclusion criteria: Eligible participants will be recruited from different outpatient clinics in Kazakhstan located in the different regions (western, eastern, northern, southern, and central parts) of the country, and must meet the following inclusion criteria: (1) age - women 18 years and older; (2) Intact uterine cervix (no prior total hysterectomy or trachelectomy); (3) ability to understand and answer questions/surveys in Kazakh, Russian or English.

Exclusion criteria: patients who are (1) younger than 18 years old, (2) women after total hysterectomy (or other surgery, when the uterine cervix is removed), (3) pregnant women, and (4) those who are not able to answer questions in Kazakh, Russian or English will be excluded.

Recruitment process. The recruitment will be done via trained and experienced outpatient gynecologists. After a careful explanation of the study's aims, all women who agreed to participate will be recruited and asked to sign an informed consent form. Further, they will (1) undergo a cervical sampling performed by the gynecologist ("gold standard" sampling), and (2) all women recruited into the study will be provided with different self-sampling kits (Evalyn Brush and Copan self-sampling swab, or Evalyn Brush and BGI Sentis HPV card) and written (picture-based) instruction to use the sampling kits. A patient will have to perform a self-sample based on the instruction and return the kits to the provider.

Sample size. We used the following parameters when estimating the required sample size: alpha = 0.05, sensitivity = 50%, accuracy estimate at 0.05%, and HPV prevalence at 40% [18]. Using the formula for sample size estimation in diagnostic studies [51], we calculated 961 participants, rounding them to 1,000 required sample size. Our goal is to survey 1000 patients to determine the acceptability of the method of self-collection of smears for HPV. With an estimated population the different regions of the country - Astana (1.000.000), Aktobe city (350.000), Almaty (around 2.000.000) - the goal to collect 1000 samples will be achieved. For this purpose, three types of HPV self-sampling kits (Evalyn Brush, Copan self-sampling swab, and BGI Sentis HPV card) will be utilized and compared.

HPV self-sampling kits. For the project purposes different types of self-sampling kits will be used - Evaline Brush, Copan self-sampling swab, the BGI company HPV self-sampling kit.

1. Evalyn Brush (https://www.roversmedicaldevices.com/cell-sampling-devices/evalyn-brush/). The Evalyn® Brush is a reliable self-sampling device for screening for the HPV.
2. Copan Self Vaginal FLOQSwabs (https://www.copangroup.com/product-ranges/self-floqswabs/) is a tube with a cotton swab. It is a comfortable device supporting women taking part in HPV and STI screening campaigns.
3. BGI Sentis HPV self-sampling kit (https://www.bgi.com/global/molecular-genetics/sentis-oncology/bgi-sentistm-hpv-test/). BGI company had established the worldwide first "communi-ty-based screening model using self-sampling HPV test as primary screening".

Surveys Women who agreed to participate in the study and perform HPV self-sampling will be asked to fill two types of questionnaires: 1) patients' socio-demographic (age, education, residence, income) and clinical data (age at menarche, number of children, gynecological and non-gynecological conditions in the past medical history, etc.); 2) and survey to assess acceptability of HPV self-sampling and different self-sampling kits.

The second questionnaire will be filled out by the participants and was adapted from previous studies. The patient questionnaire consists of 17 items (4 items to respond to before self-sampling and 13 - after) and will be used to understand patients' attitudes and acceptability of the HPV self-sampling kit. The survey will be conducted in Kazakh and Russian (or English) languages depending on the preferences of the participants.

To avoid bias, the study participants will not receive any material compensation for participation in the project.

Statistical analyses Ones the HPV testing results and questionnaires collected, statistical analysis will be performed. Statistical analyses will be performed using StataMP 16 (Stata Statistical Software: Release 16. College Station, TX: StataCorp LLC.). To validate self-sampling HPV kits, we will calculate sensitivity, specificity, positive and negative predictive values for each self-sampling HPV kit against the "gold standard" test. In univariate analysis, categorical variables will be expressed as absolute and relative frequencies, while continuous variables will be presented as means and standard deviations. To investigate attitudes and experiences about self-collection of a specimen for cervical cancer screening and understand acceptability of the method, we will use various bivariable testing techniques such as Student t-test or Mann-Whitney U-test, Pearson χ2 or Fisher's exact tests, Kruskal-Wallis test (for multiple group comparisons). Multiple logistic regression model will be used to predict the probability of the outcome based on included variables (p<0.05 or clinically important). The predictive ability of the model will be assessed based on discrimination (AUC in ROC-curve), measure of overall performance (Nagelkerke R2), calibration and decision curve analysis in STATA or R-software.

Ethical consideration The study protocol was approved by the Nazarbayev University Research Ethics Committee (NUIREC); Protocol of approval #621/03102022 (21.10.2022), "Cervical Cancer Screening Using Self-sampling Approach: Validation of Human Papillomavirus Self-sampling Kits Among Kazakhstani Women". This ethical approval was extended in 2024 until October 2025 and is subject to annual renewal.

This study will take place at Nazarbayev University School of Medicine (NUSOM) and different gynecologic hospitals/clinics across Kazakhstan. This research will include patients' self-reported clinical data questionnaire and survey to identify attitudes towards self-sampling and its acceptability. All documents related to the study (application IREC, informed consent forms, and questionnaires) were submitted to NU IREC. Informed consent will be obtained from each subject; all the documents, samples collected and results will be kept confidential. The research team will follow the principles of research ethics, in particular, preventing the fabrication of scientific data, and scientific fraud, which can lead to distortion of scientific data, plagiarism, and scientific misconduct. All patients' data (samples and surveys) will be encoded. To ensure high quality of research and obtained results, data analysis will be conducted using blind methods.

We are aware of some critical points in patient recruitment, which will be the most challenging part of the clinical research. Collaboration with the reliable team established during our previous study ("A molecular epidemiological study to determine the prevalence of oncogenic HPV strains for cervical cancer prevention in Kazakhstan", FCRGP 110119FD4528), time allocated to recruitment, specific characteristics of the population should collectively help to achieve the goals of the project.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be recruited from different outpatient clinics in Kazakhstan located in the different regions (western, eastern, northern, southern, and central parts) of the country, and must meet the following inclusion criteria:

1. age - women 18 years and older;
2. Intact uterine cervix (no prior total hysterectomy or trachelectomy);
3. ability to understand and answer questions/surveys in Kazakh, Russian or English.

Exclusion Criteria:

patients who are

1. younger than 18 years old,
2. women after total hysterectomy (or other surgery, when the uterine cervix is removed),
3. pregnant women, and
4. those who are not able to answer questions in Kazakh, Russian or English will be excluded.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants are allowed due to the nature of the study
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-sampling device acceptance | 18 months
  To assess acceptance of self-sampling modality for cervical cancer screening in Kazakhstan, various self-sampling devises will be tested:
  1. Evalyn Brush (https://www.roversmedicaldevices.com/cell-sampling-devices/evalyn-brush/).
  2. Copan Self Vaginal FLOQSwabs (https://www.copangroup.com/product-ranges/self-floqswabs/) is a tube with a cotton swab.
  3. BGI Sentis HPV self-sampling kit (https://www.bgi.com/global/molecular-genetics/sentis-oncology/bgi-sentistm-hpv-test/).
  These self-sampling kits will be distributed among the study participants who will be asked to fill surveys: : 1) patients' socio-demographic (age, education, residence, income) and clinical data (age at menarche, number of children, gynecological and non-gynecological conditions in the past medical history, etc.); 2) and survey to assess acceptability of HPV self-sampling and different self-sampling kits.

IPD SHARING:
Plan to Share IPD: No